CLINICAL TRIAL: NCT01893333
Title: The Efficacy and Safety of Nerve-sparing Radical Hysterectomy in Cervical Cancer
Acronym: NSRHCXCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSRH_Cxca
Record Dates: First submitted 2013-06-10; First posted 2013-07-09 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; nerve sparing radical hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nerve sparing radical hysterectomy group (Experimental): 1. sparing hypogastric nerve
  2. sparing pelvic splanchnic nerve ad pelvic plexus in cardinal ligament
  3. sparing distal part of hypogastric nerve and vesical branch of pelvic splanchnic nerve
  Interventions: Procedure: Nerve sparing radical hysterectomy
- Radical hysterectomy group (Active Comparator): Conventional radical hysterectomy
  Interventions: Procedure: Nerve sparing radical hysterectomy

INTERVENTIONS:
Procedure: Nerve sparing radical hysterectomy — Nerve sparing radical hysterectomy
  1. sparing hypogastric nerve
  2. sparing pelvic splanchnic nerve ad pelvic plexus in cardinal ligament
  3. sparing distal part of hypogastric nerve and vesical branch of pelvic splanchnic nerve

SUMMARY:
To develope nerve sparing radical hysterectomy for treatment of cervical cancer to minimize the complication of radical hysterectomy and to maximize quality of life and to evaluate the feasibility and efficacy by prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed cervical cancer
* FIGO stage IA2-IIA
* Diameter of tumor is less than 4cm on exam
* One of hitological type written below squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma
* Age between 18-70
* Performance status; GOG 0-1
* Normal hematological, hepatic, nephrologic function WBC ≥ 4000 cells/mm3 Platelet ≥ 100,000 /mm3 Hemoglobin ≥ 8.0 gm/dL Serum creatinin ≤ 1.3 mg/dL Serum bilirubin ≤ 1.5 mg/dL SBOT/SGPT and Alkaline phoaphatase < normal X 3
* Patient with informed consent

Exclusion creteria:

* Small cell carcinoma
* Unable to perform surgery because of severe underlying medical disease severe heart disease, congestive heart failure/severe pulmonary disease, pulmonary failure/ active bacterial infectio which needs non oral antibiotic therapy/ associated with other severe medical diseases
* Prior chemotherapy or radiotherapy
* Severe bladder funtion abnormality
* Double primary malignant tumor
* Psychiatric problems
* Pregnant or breast feeding status
* Legally unable to participate clinical trial
* When there is a Doctor's decision that patient is unable to participate clinical trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of bladder dysfunction after surgery | 5 days after the surgery
  Remove foley catheter and measure the residual urine volume Measure how long it took to be residual urine volume under 50 mL

SECONDARY OUTCOMES:
rectal & anal function after surgery | 6, 12 months after surgery
Sexual function | 6, 12 months after surgery
Quality of life | 6, 12 months after surgery
operative time | immediately after surgery
amount of bleeding in operation | immediately after surgery
frequency of blood transfusion | within 1 week after surgery
amount of blood transfusion | within 1 week after surgery
postoperative complication | within 1 month after surgery
time from surgery to return to work | within 1 month after surgery
management cost | within 1 week after surgery
size of resected parametrial tissue | immediately after surgery
2year disease free survival | 2 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea